CLINICAL TRIAL: NCT06764680
Title: Trifluridine and Tipiracil Hydrochloride Tablets, Bevacizumab and Sintilimab With/Without Involved Lesions Irradiation as 3rd- or Later-line Therapy for Advanced MSS/pMMR Colorectal Cancer: a Phase 2, Double Cohort Clinical Trial
Brief Title: Oral Chemotherapy, Targeted Therapy and Immunotherapy With/Without Radiotherapy as 3rd- or Later-line Therapy for Advanced MSS/pMMR Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, WeiWei Xiao, Prof., Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2024-585-01
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer Metastatic; Chemotherapy; Targeted Therapy; Immunotherapy; Radiotherapy, Intensity-Modulated
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- three-drug combination (Experimental): trifluorouracil tepidopyrimidine, bevacizumab, and sindilizumab
  Interventions: Drug: Trifluorouracil tepidopyrimidine; Drug: Bevacizumab; Drug: Sindilizumab
- three-drug combination and radiotherapy (Experimental): trifluorouracil tepidopyrimidine, bevacizumab, and sindilizumab combine with palliative radiotherapy of the lesions
  Interventions: Drug: Trifluorouracil tepidopyrimidine; Drug: Bevacizumab; Drug: Sindilizumab; Radiation: IMRT

INTERVENTIONS:
Drug: Trifluorouracil tepidopyrimidine — 30mg/m2. P.O. bid. d1-d5 and d15-d19. q4w
Drug: Bevacizumab — 5mg/kg. ivgtt. d1 and d15. q4w
Drug: Sindilizumab — 200mg. ivgtt. d1. q4w
Radiation: IMRT — In terms of obstruction, bleeding, compression, or pain due to a tumor that requires local treatment. IMRT was delivered to the involved lesions.
  Arms: three-drug combination and radiotherapy

SUMMARY:
The current phase 2, double cohort clinical trial was designed to determine the effectiveness of Trifluridine and Tipiracil Hydrochloride Tablets, Bevacizumab and Sintilimab with/without involved lesions irradiation as 3rd- or later-line therapy for advanced MSS/pMMR colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer ranks among the top three in terms of incidence and mortality of tumors in the world, and it is a major load on the global and China's medical and health care services. In China, about 60% of the patients are in relatively advanced stage at the time of diagnosis, and the 5-year overall survival rate is less than 15%, which is a serious threat to people's life safety. The treatment of advanced metastatic colorectal cancer which comprises of chemotherapy, mainly including oxaliplatin, irinotecan and 5-fluorouracil drugs, and target therapy, mainly including anti-EGFR and anti-vascular drugs, has led to a significant prolongation of the overall survival of patients with advanced colorectal cancer, up to about 30 months.

In terms of the chemotherapy regimens for advanced colorectal cancer, oxaliplatin and irinotecan based chemotherapy regimens are mutual first and second line, and third line and above after failure, there are some limited options available, but there are obvious limitations. Anti-VEGFR TKI-targeted therapies such as regorafenib and furaquintinib, although among the commonly available treatment options for third-line treatment of advanced colorectal cancer, have very limited efficacy rates, all less than 5%, and patients' survival time has been prolonged by only a very limited 1-2 months. Studies in the last two years have found that combining immunotherapy with an anti-VEGFR TKI can further improve efficacy, and the REGONIVO study assessed the efficacy and safety of regorafenib versus nabumab in patients with advanced colorectal cancer, and achieved an ORR of up to 36%. However, subsequent clinical studies could not achieve such favorable outcomes, and it is hypothesized that this may be related to the small percentage of liver metastases in the patients enrolled in this study. Several clinical studies have shown that anti-VEGFR TKIs combined with PD-1 monoclonal antibody have an efficacy rate of 10%-20%, which is still very limited, and more effective therapeutic strategies need to be determined.

Trifluridine-tipyrimidine is a new oral cytotoxic chemotherapy drug. Trifluridine tepipiridine consists of FTD and TPI, FTD can replace thymine into the DNA double-stranded to play an anti-tumor effect, while TPI can inhibit thymidine phosphorylase activity, prevent FTD degradation to maintain sufficient blood concentration to play a potentiating role. Bevacizumab is a recombinant humanized immunoglobulin G1 monoclonal antibody, which can effectively neutralize the vascular endothelial cell growth factor (VEGF) and inhibit its binding to the receptor, thus inhibiting its biological effects and achieving the effect of inhibiting tumor angiogenesis. Bevacizumab in combination with chemotherapy is currently used in multiple lines of treatment for advanced colorectal cancer. Trifluridine tepicillin combined with bevacizumab can appropriately improve the survival time of colorectal cancer patients, Pfeiffer et al. conducted a phase II clinical trial showed that trifluridine tepicillin combined with bevacizumab significantly prolonged the survival of the patients compared with single-agent trifluridine tepicillin, but the survival time of the combination group was still limited, with the median progression-free survival of only 4.6 months, and the median overall survival was only 9.6 months. The median overall survival was only 9.4 months, which still needs further improvement.

The most common sites of metastatic colorectal metastases are liver, lung, and bone, respectively, and some studies have found that intensive treatment of metastases improves overall survival. In surgically resected liver metastases, the 5-year overall survival rate for colorectal cancer patients ranges from 50% to 60%. However, in some cases, many patients with metastases cannot be treated with surgery due to the size and location of the tumor, and palliative radiotherapy can be used not only as an alternative to surgery, but also as a complementary treatment. In addition, radiotherapy can eliminate residual lesions or positive margins after surgical resection and reduce the risk of local recurrence. Besides, radiotherapy has been shown to activate the immune system, and the immunomodulation by radiotherapy is related to the dose and segmentation. In vitro studies have shown that a single high dose (10Gy) is more likely to induce cellular DNA damage and produce tumor neoantigens, and to activate the rapamycin pathway, which accelerates protein degradation and presentation, than a single low dose of radiation. High-dose exposures tend to induce the expression or release of immunogenic cell death-associated molecules. Compared with single high-dose irradiation, multiple high-divided radiotherapy is more likely to induce systemic immune effects. Several animal studies have found that high-divided irradiation of 8Gy×3F, 6Gy×5F, 5Gy×3F and 5Gy×4F is more likely to induce tumor growth inhibition in non-irradiated areas. Analysis of tumor-draining lymph nodes revealed that 5Gy×3F was more likely to stimulate immune cell activation than 15Gy×1F. Given that T cells are very sensitive to radiation, large fractionated radiotherapy is more favorable for lymphocyte protection.

In summary, for patients with advanced colorectal cancer, this study proposes to use a three-drug combination of trifluorouracil tepidopyrimidine, bevacizumab, and sindilizumab. For patients who meet the indications for radiotherapy, this study proposes to combine palliative radiotherapy of the lesion with the three-drug treatment. And to explore the efficacy and safety of the new combination regimen in this type of patients.

ELIGIBILITY:
Inclusion Criteria:

1. patients with advanced colorectal adenocarcinoma of MSS/pMMR confirmed by histologic or cytologic diagnosis;
2. aged 18 years and older;
3. have a quality of life score of 0-1 according to the Eastern Cooperative Oncology Group (ECOG);
4. can take oral medications;
5. expected survival ≥ 3 months;
6. progressed after standard second-line or more than second-line therapy (received oxaliplatin, irinotecan, and fluorouracil analogs);
7. have a measurable target lesion according to RECIST v1.1 evaluation criteria;
8. have a number of recurrent metastatic organs ≤ 2 for all measurable lesions, a maximum diameter of recurrent metastatic lesions ≤ 5 cm, and a total number of recurrent metastatic lesions ≤ 10;
9. agree to provide previously stored tumor tissue specimens or perform biopsies to collect tumor lesion tissue for biomarker analysis
10. have chest, abdomen and pelvis CT or whole body PET-CT results within 4 weeks before enrollment;
11. no ascites;
12. having adequate major organ function, electrocardiogram, blood, biochemistry and other basic tests to exclude contraindications to chemotherapy and radiotherapy;
13. hemoglobin >8g/L, platelets ≥100×10^9/L, neutrophils ≥1.5×10^9/L
14. for patients with liver metastases, aminotransferases and bilirubin < 5 times the upper limit of normal;
15. for patients without liver metastases, aminotransferases and bilirubin should be <2.5 times the upper limit of normal.
16. women of childbearing age must have a negative pregnancy test and conscientiously observe contraceptive measures;
17. prior systemic systemic therapy and radiation therapy for other lesions are allowed;
18. in case of discomfort such as obstruction, bleeding, compression and pain caused by the tumor, the clinical situation that local treatment may benefit the patient may be discussed between the doctor and the patient as to whether radiation therapy is to be taken;
19. if radiotherapy is required, the patient can be kept in a fixed position during radiotherapy;
20. If SABR treatment is required, the patient can tolerate the physical restraint of the immobilization device;
21. good control of the primary site: at least 3 months from radical treatment of the primary tumor, with no disease progression at the site of the primary site; or the primary tumor is not radically treated but, in the judgment of the investigator, there is no current disease progression and no threat to the patient's survival, and there is no indication for local therapy.

Exclusion Criteria:

1. prior application of trefluridine tepidopyrimidine;
2. prior application of PD-1 or PD-L1 monoclonal antibody;
3. extensive bone metastases;
4. extensive peritoneal metastases;
5. malignant hydrothorax and ascites;
6. clinical or imaging signs of spinal cord compression, or dural sac tumor visible on MRI within 2 mm of the spinal cord. If surgically resectable, it may be enrolled, but a maximum of 3 surgical sites are allowed;
7. unstable brain metastases with clinical signs or imaging evidence that require surgical decompression;
8. brainstem metastases;
9. metastatic lesions invading any of the following structures: gastrointestinal tract (including esophagus, stomach, small intestine, large intestine), skin. Includes extensive/poppy metastatic disease (e.g., brain, bone, lung, liver), or other sites where an adequate dose of irradiation could not be given (e.g., lymphovascular dissemination, malignant pleural and abdominal fluid, molluscum contagiosum metastases);
10. multiple intracranial metastases only;
11. pregnant or lactating females;
12. no reliable contraception during the reproductive period
13. patients with a known history of hypersensitivity to any of the study drugs, analogs, or excipients;
14. patients at risk of gastrointestinal hemorrhage or gastrointestinal obstruction;
15. patients with a history of thromboembolism, with the exception of thrombosis caused by PICCs or infusion ports
16. patients with difficult-to-control hypertension (systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥90 mmHg after optimal antihypertensive treatment);
17. patients with contraindications to treatment such as other chronic diseases;
18. Patients with active infections;
19. patients with a pre-existing condition of immunotherapy-associated myocarditis, pneumonia, colitis, hepatitis, or nephritis who, in the judgment of the investigator, are at greater risk for reuse of immunotherapy;
20. patients with existing toxic side effects ≥ grade 2 due to prior therapy according to NCI CTCAE version 5.0 (except for alopecia, hyperpigmentation, etc.);
21. severe medical comorbidities that preclude radiotherapy, including interstitial lung disease with current metastases requiring radiotherapy to the lungs, Crohn's disease requiring radiotherapy to the gastrointestinal tract, or connective tissue disease such as lupus erythematosus or scleroderma;
22. there is an overlap between the current radiation field and the field of prior radiotherapy. It may be permissible to have had prior radiation therapy as long as the fusion cumulative dose meets the dose limits. For this case, request that the dose be accrued in accordance with the BED and discuss with the PI whether this can be performed;
23. prior systemic nuclide therapy, such as Radium-223 or Lutetium-177);
24. other circumstances that the investigator determines are not appropriate for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Baseline, 6-8 weeks after treatment complete
  Objective response rate (ORR) was defined as the percentage of CR+PR among the patients who could be evaluated for efficacy.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Baseline, 6-8 weeks after treatment complete
  Disease control rate (DCR) was defined as the percentage of CR+PR+SD among the patients who could be evaluated for efficacy.
Progression-free survival (PFS) | month 6, year 1, year 2
  Progression-free survival (PFS) was calculated from the date of treatment to either the date of disease progression, death or last follow-up.
Overall survival (OS) | month 6, year 1, year 2
  Overall survival (OS) was calculated from the date of treatment to either the date of death or last follow-up.
Treatment related toxicity | Baseline, 6-8 weeks after treatment complete
  Grading of acute toxicity would be assessed according to National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Weiwei Xiao, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China